CLINICAL TRIAL: NCT00004735
Title: The Effects of Highly Active Antiretroviral Therapy (HAART) on the Recovery of Immune Function in HIV-Infected Children and Young Adults
Brief Title: The Effects of Anti-HIV Therapy on the Immune Systems of Children and Young Adults Infected With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACTG P1006; 10036 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2000-02-25; First posted 2001-08-31 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: HIV Infections
Keywords: Viral Vaccines; Drug Therapy, Combination; CD4-Positive T-Lymphocytes; Immunologic Memory; Antibody Formation; Anti-HIV Agents; Tetanus Toxoid; Hepatitis A Virus, Human; Enfuvirtide; T-20; Treatment Naive; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Tetanus; Hepatitis | interventions — Tetanus Toxoid; Hepatitis A Vaccines

INTERVENTIONS:
Biological: Tetanus toxoid
Biological: Hepatitis A Vaccine (Inactivated)

SUMMARY:
The purpose of this study is to determine the number of newly formed CD4 cells in children who have taken anti-HIV drugs. The study will also evaluate the effectiveness of the new CD4 cells in producing an immune response to hepatitis A and tetanus toxoid vaccination.

Study hypothesis: 1) Immunologic reconstitution of individuals who have less than 15% CD4 cells may or may not be associated with functional activity. 2) The functional immunologic responses to recall and newly experienced antigens may be different. 3) The functional responses to antigens delivered in vaccine format may be a function of CD4 level, viral load, or both.

DETAILED DESCRIPTION:
HIV damages the immune system by infecting CD4 cells, white blood cells that help fight infections and protect the body from disease. As CD4 cells die, the immune system becomes weak. Taking anti-HIV drugs slows the ability of the virus to multiply and kill CD4 cells. HIV infected children taking anti-HIV drugs have significant inhibition of HIV growth and significant increases in CD4 cell counts. It is not known to what extent CD4 count increases in HIV infected children translate to functional immune recovery. HIV infected children have typically demonstrated poor serological responses to routine childhood immunizations.

Participants will either begin HAART or make a change to their current HAART regimens at study entry or within 2 weeks prior to study entry. All participants will have viral load testing when they begin or change their HAART regimens. Participants will then have a second viral load test after 4 weeks. Only participants with an acceptable decrease in viral load will continue in the study.

Participants will be randomly assigned to one of two groups. Participants in Group 1 will receive tetanus toxoid immunizations (known as DTaP, DT-pediatric, or Td) at Weeks 8, 16, and 24 and hepatitis A vaccinations at Weeks 32, 40, and 48. Participants in Group 2 will receive hepatitis A vaccinations at Weeks 8, 16, and 24 and tetanus toxoid immunizations at Weeks 32, 40, and 48. Participants will have a physical exam and blood tests at study entry and at Weeks 4, 8, 12, 16, 24, 28, 32, 36, 40, 48, 52, 76, and 100.

As of May 2005, participants will have the option to receive an additional hepatitis A vaccination booster. Those who consent and have not reached Week 100 of the study will receive a booster vaccination at Week 100, with a final follow-up visit occuring at Week 104. Those participants who do not consent will not receive the hepatitis A vaccination booster and will have their last follow-up visit at Week 100.

ELIGIBILITY:
Inclusion Criteria

* HIV infected
* CD4 percentage less than 15%
* Beginning an anti-HIV drug regimen (HAART) that includes at least 3 drugs. Two of the drugs must be new to the patient. One of the new drugs must be a protease inhibitor or a nonnucleoside reverse transcriptase inhibitor (NNRTI). As of May 2005, patients who have previously taken NNRTIs will have the option of taking Fuzeon as an alternative component of their HAART regimen
* Consent of parent or legal guardian
* As of May 2005, females who become pregnant during the study can continue to participate as long as they become pregnant after receiving all vaccinations

Exclusion Criteria

* Active opportunistic (AIDS-related) or bacterial infection
* Cancer
* Immunity to hepatitis A
* Severe drug toxicity
* Previous severe or allergic reaction to tetanus vaccine
* Taking IVIG, IL-2, or other drugs which affect the immune system
* Taking hydroxyurea
* Pregnancy at screening visit
* Pregnancy before all vaccinations have been administered

Ages: 2 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2000-02; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
A stimulation index of 3 or greater on at least 2 occasions to tetanus
positive serologic response to hepatitis A
four-fold increase over baseline in antibody titers for tetanus

SECONDARY OUTCOMES:
A stimulation index of 3 or greater on at least 2 occasions to hepatitis A and Candida
increase in CD4 cell percentage by 10% and absolute CD4 number by 150 cells/ml
development of any adverse events of Grade 3 or higher attributable to vaccination

CONTACTS AND LOCATIONS:
Overall Officials: William Borkowsky, MD, Study Chair — NYU Langone Health; Mona Rigaud, MD, MPH, Study Chair — NYU Langone Health
Locations (27):
- United States (25):
  - UAB, Dept. of Ped., Div. of Infectious Diseases, Birmingham, Alabama
  - Usc La Nichd Crs, Alhambra, California
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Children's National Med. Ctr., ACTU, Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - South Florida CDTC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Univ. of Florida College of Medicine-Dept of Peds, Div. of Immunology, Infectious Diseases & Allergy, Gainesville, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - USF - Tampa NICHD CRS, Tampa, Florida
  - Chicago Children's CRS, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Schneider Children's Hosp., Div. of Infectious Diseases, New Hyde Park, New York
  - Nyu Ny Nichd Crs, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - Strong Memorial Hospital Rochester NY NICHD CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - UW School of Medicine - CHRMC, Seattle, Washington
- Puerto Rico (2):
  - San Juan City Hosp. PR NICHD CRS, San Juan
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan

REFERENCES:
- [Background] Melvin AJ, Mohan KM. Response to immunization with measles, tetanus, and Haemophilus influenzae type b vaccines in children who have human immunodeficiency virus type 1 infection and are treated with highly active antiretroviral therapy. Pediatrics. 2003 Jun;111(6 Pt 1):e641-4. doi: 10.1542/peds.111.6.e641. PMID 12777579
- [Result] Rigaud M, Borkowsky W, Muresan P, Weinberg A, Larussa P, Fenton T, Read JS, Jean-Philippe P, Fergusson E, Zimmer B, Smith D, Kraimer J; Pediatrics AIDS Clinical Trials Group P1006 Team. Impaired immunity to recall antigens and neoantigens in severely immunocompromised children and adolescents during the first year of effective highly active antiretroviral therapy. J Infect Dis. 2008 Oct 15;198(8):1123-30. doi: 10.1086/592050. PMID 18752430